CLINICAL TRIAL: NCT06715839
Title: Development and Clinical Translation of immunoPET Imaging Probes for Digestive System Carcinoma
Brief Title: Target-specific immunoPET Imaging of Digestive System Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KY2024-107-C
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Malignancy; Digestive Cancer; Digestive System Neoplasm; Digestive System Carcinoma; Digestive System Cancer; Liver Cancer; Stomach Cancer; Colon Cancer; Rectum Cancer; Pancreatic Cancer; Esophagus Cancer; Gallbladder Carcinoma; Small Intestine Cancer; Appendix Cancer; Bile Duct Carcinoma
Keywords: human epidermal growth factor receptor 2 (HER2); Trophoblast cell surface antigen 2 (TROP2); Glypican-3 (GPC3); Glycoprotein A33 (gpA33); Nectin cell adhesion molecule-4 (Nectin-4)
MeSH Terms: conditions — Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Liver Neoplasms; Stomach Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Pancreatic Neoplasms; Esophageal Neoplasms; Gallbladder Neoplasms; Appendiceal Neoplasms; Bile Duct Neoplasms; Simpson-Golabi-Behmel syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ImmunoPET imaging in patients with digestive system carcinoma (Experimental): Enrolled patients will undergo a targeted-specific immunoPET/CT scanning.
  Interventions: Drug: [68Ga]Ga-DOTA-H2D3; Drug: [18F]F-RESCA-RB14; Drug: [68Ga]Ga-NOTA-T4; Drug: [18F]F-RESCA-T4; Drug: [68Ga]Ga-NOTA-G5; Drug: [18F]F-RESCA-G5; Drug: [68Ga]Ga-NOTA-WWH347; Drug: [18F]F-RESCA-WWH347; Drug: [68Ga]Ga-NOTA-RND20; Drug: [18F]F-RESCA-RND20

INTERVENTIONS:
Drug: [68Ga]Ga-DOTA-H2D3 — Enrolled patients (especially those with gastric cancer) will receive 0.05-0.1 mCi/kg of a HER2-targeted probe ([68Ga]Ga-DOTA-H2D3). ImmunoPET/CT imaging will be acquired 1-2 hours after [68Ga]Ga-DOTA-H2D3 injection.
  Other Names: [68Ga]Ga-H2D3
Drug: [18F]F-RESCA-RB14 — Enrolled patients (especially those with gastric cancer) will receive 0.05-0.1 mCi/kg of a HER2-targeted probe ([18F]F-RESCA-RB14). ImmunoPET/CT imaging will be acquired 1-2 hours after [18F]F-RESCA-RB14 injection.
  Other Names: [18F]F-RB14
Drug: [68Ga]Ga-NOTA-T4 — Enrolled patients (especially those with gastric cancer/pancreatic cancer) will receive 0.05-0.1 mCi/kg of a Trop2-targeted probe ([68Ga]Ga-NOTA-T4). ImmunoPET/CT imaging will be acquired 1-2 hours after [68Ga]Ga-NOTA-T4 injection.
  Other Names: [68Ga]Ga-T4
Drug: [18F]F-RESCA-T4 — Enrolled patients (especially those with gastric cancer/pancreatic cancer) will receive 0.05-0.1 mCi/kg of a Trop2-targeted probe ([18F]F-RESCA-T4). ImmunoPET/CT imaging will be acquired 1-2 hours after [18F]F-RESCA-T4 injection.
  Other Names: [18F]F-T4
Drug: [68Ga]Ga-NOTA-G5 — Enrolled patients (especially those with hepatocellular carcinoma) will receive 0.05-0.1 mCi/kg of a GPC3-targeted probe ([68Ga]Ga-NOTA-G5). ImmunoPET/CT imaging will be acquired 1-2 hours after [68Ga]Ga-NOTA-G5 injection.
  Other Names: [68Ga]Ga-G5
Drug: [18F]F-RESCA-G5 — Enrolled patients (especially those with hepatocellular carcinoma) will receive 0.05-0.1 mCi/kg of a GPC3-targeted probe ([18F]F-RESCA-G5). ImmunoPET/CT imaging will be acquired 1-2 hours after [18F]F-RESCA-G5 injection.
  Other Names: [18F]F-G5
Drug: [68Ga]Ga-NOTA-WWH347 — Enrolled patients (especially those with colorectal cancer) will receive 0.05-0.1 mCi/kg of a GPA33-targeted probe ([68Ga]Ga-NOTA-WWH347). ImmunoPET/CT imaging will be acquired 1-2 hours after [68Ga]Ga-NOTA-WWH347 injection.
  Other Names: [68Ga]Ga-WWH347
Drug: [18F]F-RESCA-WWH347 — Enrolled patients (especially those with colorectal cancer) will receive 0.05-0.1 mCi/kg of a GPA33-targeted probe ([18F]F-RESCA-WWH347). ImmunoPET/CT imaging will be acquired 1-2 hours after [18F]F-RESCA-WWH347 injection.
  Other Names: [18F]F-WWH347
Drug: [68Ga]Ga-NOTA-RND20 — Enrolled patients will receive 0.05-0.1 mCi/kg of a Nectin-4-targeted probe ([68Ga]Ga-NOTA-RND20). ImmunoPET/CT imaging will be acquired 1-2 hours after [68Ga]Ga-NOTA-RND20 injection.
  Other Names: [68Ga]Ga-RND20
Drug: [18F]F-RESCA-RND20 — Enrolled patients will receive 0.05-0.1 mCi/kg of a Nectin-4-targeted probe ([18F]F-RESCA-RND20). ImmunoPET/CT imaging will be acquired 1-2 hours after [18F]F-RESCA-RND20 injection.
  Other Names: [18F]F-RND20

SUMMARY:
The aim of this study is to establish and optimize the target-specific PET/CT imaging method, and its physiological and pathological distribution characteristics, on the basis of which the diagnostic efficacy of the above imaging agents in digestive system malignant tumors will be evaluated.

DETAILED DESCRIPTION:
Enrolled patients will undergo whole-body PET/CT scans at 1 hours after tracer injection(0.05-0.1 mCi/kg). Uptake of above imaging agents in tumor and normal organs/tissues will be scored visually and quantitatively.

Tumor uptake will be quantified by the maximum standard uptake value (SUVmax). The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and accuracy will be calculated to evaluate the diagnostic efficacy. The correlation between lesion uptake and protein expression level determined by immunohistochemistry staining will be further analyzed. The exploration endpoint will be the imaging feasibility and preliminary diagnostic value of the above tracers.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years old and of either sex；
2. Histologically confirmed diagnosis of digestive system carcinoma or suspected digestive system carcinoma by diagnostic imaging;
3. Capable of giving signed informed consent, including compliance with the requirements and restrictions listed in the informed consent form (ICF) and this protocol.

Exclusion Criteria:

1. Pregnancy；
2. Severe hepatic and renal insufficiency;
3. History of serious surgery in the last month;
4. Allergic to antibody or single-domain antibody radiopharmaceuticals.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Biodistribution | 1 day from injection of the tracers
  Measurement of the overall biodistribution of above tracers in normal tissues and organs.
Standardized uptake value (SUV) | 1 day from injection of the tracers
  Standardized uptake value (SUV) of above tracers in the included subjects' primary and/or metastatic lesions.
Radiation dosimetry | 1 day from injection of the tracers
  Measurement of absorbed radiation doses (Gy/MBq) to tissues/organs, tumor(s), and whole body (Sv/MBq). Dynamic imaging within one hour will be acquired for the purpose.
Diagnostic value in patients with digestive system malignancy | 30 days
  Systematic evaluation of these parameters will elucidate the pharmacokinetics, pharmacodynamics and, more importantly, the clinical value of these target-specific tracers in patients with malignancies of the digestive system.
The correlation between the expression of specific target and tracer uptake value | 60 days
  The Standardized uptake value (SUV) will be calculated, and the correlation between pathological results and tumor uptake of these tracers will be analyzed.

SECONDARY OUTCOMES:
Predictive value of these tracers in the course of combined immunotherapies and targeted therapies | 3-6 months
  Baseline and follow-up immunoPET imaging in combined immunotherapies and targeted therapies (four to eight cycles) will be investigated in this setting to determine the value of the immunoPET imaging in predicting or evaluating treatment responses.
Target-specific PET/CT in changing clinical decision-making for patients with digestive system malignancy | 3-6 months
  After analyzing the imaging parameters and diagnostic/predictive value of these target-specific tracers, we will also investigate how clinical use of these tracers changes clinical decision-making for patients with malignant tumors of the digestive system. Joint efforts from nuclear medicine physicians, surgeons, oncologists, and pathologists will draw solid conclusions from the imaging and clinical information.

CONTACTS AND LOCATIONS:
Overall Officials: Weijun Wei, Study Chair — Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China